CLINICAL TRIAL: NCT05507684
Title: RECETAS (Re-Imagining Environments for Connection and Engagement: Testing Actions for Social Prescribing in Natural Spaces) in Helsinki
Brief Title: Effects of Nature-based Group Intervention on Quality-of-life in Lonely Older People Living in Assisted Living Facities
Acronym: RECETAS
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Helsinki (Other)
Collaborators: Barcelona Institute of Global Health (Unknown); Helsinki City Older People's Services (Unknown); The Finnish Association for the Welfare of Older People (Unknown)
Responsible Party: Principal Investigator, Kaisu Pitkala, PhD, Professor emerita, University of Helsinki
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 945095 HEL
Record Dates: First submitted 2022-08-12; First posted 2022-08-19 (Actual); Last update posted 2025-02-28 (Actual); Status verified 2025-02

CONDITIONS: Loneliness
Keywords: Loneliness, nature activities, group intervention, socialization

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Nature-based social prescribing group intervention (Experimental): Groups of 5-12 persons will formed from one assisted living facility. All of them will undergo an individual interview to assess their wishes for the nature-based activities.
  Participants meet in a closed group 9 times for once a week for 10 weeks. All 2-4 hour sessions will include nature-based activities and mutual discussions about the experiences of nature and loneliness.
  2 professionals will facilitate and observe the group more thoroughly, give feedback to each other, and make use of group dynamics. They write diaries on each session and receive feedback from their trainers. The groups are objective oriented (aiming to alleviate loneliness, to improve participants' self-efficacy), client oriented and aim with favorable group dynamics to mature, self-directing group in which the participants have made friends with each other and want meet with each other without the facilitators after the official group intervention is over.
  Interventions: Other: Nature-based social prescribing group intervention
- Control (No Intervention): The control arm will receive individually usual care in assisted living facility (e.g. the existing social prescription as available) Usual care is the appropriate comparison rather than a placebo for complex interventions.

INTERVENTIONS:
Other: Nature-based social prescribing group intervention — Groups of 5-12 persons will formed from one assisted living facility. All of them will undergo an individual interview to assess their wishes for the nature-based activities.
  Participants meet in a closed group for 9 times once a week for 10 weeks. All 2-4 hour sessions will include nature-based activities and mutual discussions about the experiences of nature and loneliness.
  2 professionals will facilitate and observe the group more thoroughly, give feedback to each other, and make use of group dynamics. They write diaries on each session and receive feedback from their trainers. The groups are objective oriented (aiming to alleviate loneliness, to improve participants' self-efficacy), client oriented and aim with favorable group dynamics to mature, self-directing group in which the participants have made friends with each other and want meet with each other without the facilitators after the official group intervention is over.
  Arms: Nature-based social prescribing group intervention

SUMMARY:
RECETAS (Re-imagining Environments for Connection and Engagement:

Testing Actions for Social Prescribing in Natural Spaces) is a worldwide project (H2020 No 945095) that addresses loneliness and the role of nature-based social intervention (NBSI) to alleviate it. Definitions: Loneliness is the perception of feeling alone, even if surrounded by people. Social prescription is a non-medical community referral approach to connect individuals with community resources to support wellbeing. Nature-based social intervention (NBSI) is a structured therapeutic groupbased social intervention that specifically include access to nature as a main component. Nature-based experiences may facilitate dynamic processes of social interactions and it can reduce feelings of loneliness.

Hypothesis: NBSI in vulnerable people suffering from loneliness is more effective than usual social and health care on improving their health-related quality of life and alleviating loneliness during 3-,6- and 12-months follow up.

Objectives: This trial aims to assess the effectiveness and to explore the processes and perceived impacts of NBSI in vulnerable people suffering from loneliness in the assisted living facilities in Helsinki. In Helsinki, the main objective is to assess the effectiveness of a 10-week NBSI (RCT) in vulnerable people suffering from loneliness on changes of their health-related quality of life (HRQOL) and loneliness compared to usual social and health care at end of intervention, and at 6-,and 12- months post-randomization.

Methods: The study design is a randomized controlled trial (RCT). The RCT will include also a process evaluation, a qualitative study and a Health Economics evaluation. Therefore, the RCT will use a mixed-method approach collecting quantitative information to assess the main outcomes and qualitative methods to explore lived experiences of participants and professionals.

The recruitment will be performed screening residents in Helsinki assisted living facilities by a survey. A total of 316 participants will be randomly allocated in two groups (c.158 each) after baseline assessments: intervention and control. Participants will sign the informed consent. The intervention is a group-based, multicomponent, behaviorally based complex intervention that requires a specific training to prepare professionals as facilitators. It is based on the "Circle of Friends" methodology.

DETAILED DESCRIPTION:
RECETAS (Re-imagining Environments for Connection and Engagement:

Testing Actions for Social Prescribing in Natural Spaces) is a worldwide project that addresses loneliness and the role of nature-based social intervention (NBSI) to alleviate it. This project has received funding from tte European Union's Horizon 2020 research and innovation under grant agreement No 945094. more information at: https://recetasproject.eu Background: Loneliness is the perception of feeling alone, even if surrounded by people. It is a growing public health concern due to its impact on morbidity and mortality even in old age, being as dangerous as smoking or obesity: it reduces people's lifespan, and it is associated with increased use of health and social services and it impairs people's quality-of-life. In Europe, 30 million European adults frequently felt lonely. Social prescription is a non-medical community referral approach to connect individuals with community resources to support wellbeing. Nature-based social intervention (NBSI) is a structured therapeutic group-based social intervention that specifically include access to nature as a main component. Nature-based experiences can facilitate dynamic processes of social interactions and it can reduce feelings of loneliness.

Justification: NBSI in urban areas may improve health and mental well-being and reduce loneliness. Investments in nature-based solutions and green infrastructure can be harnessed for health and wellbeing even in times of health emergencies (covid-19). NBSI offers a novel socio-environmental innovation to reduce loneliness by creating the social and technological infrastructure needed to support social and community cohesion.

Hypothesis: NBSI in vulnerable older people in assisted living facilities suffering from loneliness is more effective than usual social and health care on improving their quality of life and alleviating loneliness during 3-,6- and 12-months follow up.

Objectives: The study aims to assess the effectiveness and to explore the processes and perceived impacts of NBSI in vulnerable older people in assisted living facilities suffering from loneliness in the area of Helsinki. The main objective is to assess the effectiveness of a 10-week NBSI (RCT) in vulnerable people suffering from loneliness on the changes of loneliness and health-related quality of life compared to usual social and health care at 3-, 6-, and 12- months post-randomization.

Methods: The study design is a randomized controlled trial (RCT). The RCT will also include a process evaluation, a qualitative study and a health economics evaluation.

Therefore, overall, the RCT will use a mixed-method approach collecting quantitative information to assess the main outcomes and qualitative methods to explore lived experiences of participants and professionals. The recruitment will be performed by screening residents in Helsinki assisted living facilities by a survey inclusing 1500 residents. Inclusion criteria will be age 65+ years, suffering from loneliness, living permanently in assisted living facility, being voluntary to participate, having Minimental Examination at least 15 point (not being moderately-severly cognitively impaired), being able to move independently with or without assisting devices, sufficient sight and hearing and not having a seirous illnes with a prognosis than 6 months. A total of 316 participants will be randomly allocated in two groups (c.158 each) after baseline assessments: intervention and control. Participants will sign the informed consent. The intervention is a group-based, multicomponent, behaviorally based complex intervention that requires a specific training to prepare professionals as facilitators. It is based on the "Circle of Friends" methodology developed in Helsinki University. Participants in the intervention arm meet in closed groups including 5-12 participants once a week for 9 times. The group activities include nature-based activities and discussions on them and participants' loneliness. The groups facilitators will use group dynamics to facilitate participants' mutual interaction and to support their self-efficacy. Control group participants will receive usual care, and a list of nature-based resources available in their area.

Main outcome measures will be changes in loneliness by De Jong Gierveld Loneliness scale and health-related quality-of-life by 15D measure. Secondary measures will be changes in wellbeing (Psychological Wellbeing scale), EuroQual 5D-5L, cognition (Minimental State examination, Clock-drawing test, verbal fluency), walking speed and frailty (Physical frailty), self efficacy (Generalized Self-Efficacy scale), sleep quality, attachment ot neighbourhood (12 Neighborhood Assessment Scale), and relationship with nature (NR-6). THe use of health and social services will be collected from central records and health economic analyses performed.

ELIGIBILITY:
Inclusion Criteria:

* Age at least 55 years
* Suffers from loneliness at least sometimes
* lives permanently in assisted living facility
* is voluntary to participate
* has Minimental Examination at least 15 points or CPS <5 (not being moderately-severly cognitively impaired)
* is able to move independently or dependently with or without assisting devices
* sufficient sight and hearing to participate in group activities

Exclusion Criteria:

having a serious illness with a prognosis less than 6 months.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 316 (Estimated)
Dates: Start 2023-02-21 (Actual); Primary Completion 2025-01-28 (Actual); Study Completion 2026-02-28 (Estimated)

PRIMARY OUTCOMES:
Change in health related quality of life | From baseline to 3months, 6months, 12 months
  15D health-related quality of life instrument. Minimum 0 (worst) and maximum 1 (best). 15D will be used as an index ( 0 to 1) and the changes in various 15 dimensions will also be explored.
Change in loneliness | From baseline to 3months, 6months, 12 months
  Modified De Jong Gierveld Loneliness Scale as a continuous scale (minimum 11 (best) and maximum 55 (worst))

SECONDARY OUTCOMES:
Change in Psychological Wellbeing | From baseline to 3months, 6months, 12 months
  Psychological Wellbeing Scale by Routasalo et al. 2009 (Minimum 0 (worst) and maximum 1 (best).
Change in executive function | From baseline to 3months, 6months, 12 months
  Clock Drawing test (Minimum 0 (worst) and maximum 6 (best).
Change in cognition | From baseline to 3months, 6months, 12 months
  Verbal Fluency (Minimum 0 (worst) and maximum >30 (best)).
Minimental State Examination | Only baseline
Change in self Efficacy | From baseline to 3months
  Generalized Self-Efficacy scale by Schwarzer & Jerusalem 1995
Change in frailty phenotype | Only baseline
  Physical frailty
Change in blood pressure | From baseline to 3months and 12 months
  Blood pressure
Change in sleep quality | From baseline to 3months, 6months, 12 months
  One item questions
Change in attachment to neighbourhood | From baseline to 3months
  Neighborhood Assessment Scale
Change in relationship with nature | From baseline to 3months
  Questions related to nature attitudes
Use of health and social services | during 12 months from baseline
  Use of health and social services retrieved from registers
Health economic analyses (costs of health services with EQ5D-5L) | During 12 months (3mo, 6mo, 12mo)
  EuroQOL 5D-5L
Change in social relationships | From baseline to 3months, 6months, 12 months
  Number of new friends, continuation of group activity, satisfaction with relationships
Repeated wellbeing before, during and after the intervention | Baseline, during the intervention and at 3 months
  4 items related to psychological and physical wellbeing
Repeated short measure of wellbeing | Baseline, during the intervention and at 3 months
  4 items related to psychological and physical wellbeing
Satisfaction with social relationships | Baseline, 3 months
  Items on social relationships and social activity
Number and time spent on outdoor activities | 3 months from baseline
  Number of outdoor activities and time spent there during the intervention

OTHER OUTCOMES:
Group participants' opinions | during the group and at 3 months
  Group participants' opinions about the group activities and its impact on loneliness and social relationships

CONTACTS AND LOCATIONS:
Overall Officials: Jill S Litt, PhD, Principal Investigator — Barcelona Institute for Global Health
Locations (1):
- Helsinki City assisted living facilities, Helsinki, Finland

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, CSR
Time Frame: 2022 - 2026
Access Criteria: Study protocol has been submitted to a peer reviewed journal. Clinical study report will be available in 2026.

REFERENCES:
- [Derived] Pitkala KH, Rautiainen L, Kautiainen H, Aalto UL, Kolster A, Laakkonen ML, Partonen T, Roitto HM, Puntscher S, Rochau U, Siebert U, Bartova A, Holmerova I, Coll-Planas L, Litt JS, Strandberg T, Jansson AH. Effectiveness of nature-based group intervention in loneliness and health-related quality-of-life in lonely older adults living in assisted living facilities-a randomised controlled trial. Age Ageing. 2026 Feb 1;55(2):afag009. doi: 10.1093/ageing/afag009. PMID 41638234
- [Derived] Vert C, Litt JS, Gascon M, Roque M, Maso-Aguado M, Opacin N, Garcia G, Jansson A, Cattaneo L, Bartova A, Briones-Buixassa L, Carbo A, Rautiainen LJ, Hidalgo L, Sachs A, Domenech S, Blancafort-Alias S, Holmerova I, Pitkala KH, Coll-Planas L. Evaluating the feasibility of "Friends in Nature," a complex nature-based social intervention to address loneliness and quality of life in six cities worldwide. Pilot Feasibility Stud. 2024 Nov 30;10(1):146. doi: 10.1186/s40814-024-01575-4. PMID 39616375
- [Derived] Pitkala KH, Rautiainen L, Aalto UL, Kautiainen H, Kolster A, Laakkonen ML, Partonen T, Roitto HM, Strandberg TE, Opacin N, Puntscher S, Siebert U, Coll-Planas L, Sachs AL, Litt JS, Jansson AH; RECETAS project. Participants' baseline characteristics and feedback of the nature-based social intervention "friends in nature" among lonely older adults in assisted living facilities in finland: a randomised controlled trial of the RECETAS EU-project. BMC Geriatr. 2024 Oct 7;24(1):812. doi: 10.1186/s12877-024-05408-0. PMID 39375627
- [Derived] Coll-Planas L, Carbo-Cardena A, Jansson A, Dostalova V, Bartova A, Rautiainen L, Kolster A, Maso-Aguado M, Briones-Buixassa L, Blancafort-Alias S, Roque-Figuls M, Sachs AL, Casajuana C, Siebert U, Rochau U, Puntscher S, Holmerova I, Pitkala KH, Litt JS. Nature-based social interventions to address loneliness among vulnerable populations: a common study protocol for three related randomized controlled trials in Barcelona, Helsinki, and Prague within the RECETAS European project. BMC Public Health. 2024 Jan 13;24(1):172. doi: 10.1186/s12889-023-17547-x. PMID 38218784